CLINICAL TRIAL: NCT06605157
Title: Pilot Randomized Clinical Trial of A Multimodal Music Therapy Intervention for Engaging Persons With Severe Dementia (AMUSED)
Brief Title: A Multimodal Music Therapy Intervention for Engaging Persons With Severe Dementia
Acronym: AMUSED
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Alaine E Hernandez, PhD (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor-Investigator, Alaine E Hernandez, PhD, Assistant Professor of Music Therapy, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 94750; P30AG072946 (NIH)
Record Dates: First submitted 2024-09-06; First posted 2024-09-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Dementia Severe
Keywords: Music Therapy; Evidence-based practice; Behavioral symptoms; Speech; Language; Artificial intelligence
MeSH Terms: conditions — Behavioral Symptoms; Speech; Language

STUDY DESIGN:
Intervention Model Description: To prevent cross-contamination, a research team member will randomize facilities as clusters (N=8) 1:1 to either the music or the reading intervention using a random number table. Opting for four clusters per arm will enable the researchers to estimate cluster effects and evaluate delivery across different care structures. The researchers will enroll at least 5 participants from each cluster/facility to provide a buffer against attrition to maintain a group of at least 3 individuals in each cluster. Delivery of both music and reading is in small groups (3-5 people).
Who Masked: Investigator
Masking Description: Participants and care providers (music therapists, reading group leaders) will not be masked; both will know what is being received (music therapy or reading). Principal investigator Reschke-Hernandez and Co-Is Schmitt and Abner will remain masked to allocation. Care staff who collect behavior data will not be masked; care staff will know if the facility is receiving music therapy or reading. However, for all other outcomes, research assistants who assess participants will be masked to group assignment without knowledge of the intervention assigned to individual participants. Allocation and assignment information will be kept in a separate secure document that is not accessible to the PI or Co-Is.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Music Therapy (Experimental): Live delivery of a music therapy protocol that is designed to be led by a board-certified music therapist (MT-BC). Activity blocks are identical to the reading arm:
  * T0 Baseline measures
  * Weeks 1-4: music therapy intervention
  * T1 measures (end of week 4)
  * Weeks 5-8: music therapy intervention
  * T2 measures (end of week 8)
  * Weeks 5-8: music therapy intervention
  * T3 measures (end of week 12)
  * T4 measures 4-week-follow-up (week 16)
  Interventions: Behavioral: AMUSED
- Reading Aloud (Active Comparator): Live reading aloud of an age-appropriate book by a group leader to control for social attention and isolate the effects of music.
  Activity blocks are identical to the music therapy arm:
  * T0 Baseline measures
  * Weeks 1-4: music therapy intervention
  * T1 measures (end of week 4)
  * Weeks 5-8: music therapy intervention
  * T2 measures (end of week 8)
  * Weeks 5-8: music therapy intervention
  * T3 measures (end of week 12)
  * T4 measures 4-week-follow-up (week 16)
  Interventions: Behavioral: Reading Aloud

INTERVENTIONS:
Behavioral: AMUSED — Delivered live by a board-certified music therapist (MT-BC) 40 min 2x/week for 12 weeks (24 total sessions; 16 total hours) in small groups of 3-5 people. A Multimodal mUSic therapy intervention for Engaging persons with severe Dementia (AMUSED) uses live participant-preferred music and progressively layers singing, touch, and rhythmic instrument playing concurrent with participant behavioral responses. Follows the Clinical Practice Model for Persons with Dementia and implementation strategies that promote cognition, attention, familiarity, audibility, structure, autonomy per participants' strengths, interests, preferences, culture, and momentary responses. Each small group works with the same music therapist throughout the study.
  Arms: Music Therapy
Behavioral: Reading Aloud — Delivered live by a trained research assistant ("interventionist") 40 min 2x/week for 12 weeks (24 total sessions; 16 total hours) in small groups of 3-5 people. The interventionist will read aloud from age-appropriate books (Chicken Soup for the Golden Soul by Jack Canfield; World of Wonders by Aimee Nezhukumatathil) selected to have sufficient material for all sessions, contain short stories to accommodate for attention span and session length, and offer choice. Follows implementation strategies identical to the music therapy arm (i.e., within the Clinical Practice Model for Persons with Dementia) that promote cognition, attention, familiarity, audibility, structure, autonomy per participants' strengths, interests, preferences, culture, and momentary responses. However, no music (including musical references) is used. Each small group works with the same reading interventionist throughout the study.
  Arms: Reading Aloud

SUMMARY:
The goal of this pilot randomized clinical trial is to learn if a music therapy treatment, called AMUSED, can improve engagement and reduce behavioral symptoms in older adults with severe dementia who live in care facilities. The main questions it aims to answer are:

* Is it feasible to conduct a full-scale trial of AMUSED?
* Can investigators identify the best outcome measures to assess impact on behavioral symptoms of dementia?
* Does speech offer a useful indicator of treatment effectiveness? Researchers will compare a group-based music therapy treatment to a reading activity to learn if music therapy leads to greater improvements in behavioral symptoms and speech patterns.

Participants will:

* Participate in either music therapy (includes live music, singing, and rhythmic instrument playing) or a reading group with stories about life and nature and talk about memories.
* Attend small group sessions twice a week for 12 weeks, with each session lasting 40 minutes between lunch and dinner.
* Be observed and assessed for behavioral symptoms, cognition, and speech several times during treatment and at a 4-week follow-up.

DETAILED DESCRIPTION:
Meaningful activity has personal importance or usefulness, fosters a sense of fulfillment, and contributes to well-being, whether through cherished pastimes or goal-oriented endeavors. Persons with dementia (PWD) experience significant deficits in memory, communication, and functional abilities, which poses unique obstacles to engage in meaningful activities. When PWD lack sufficient activity, or if activities are poorly tailored to ability, PWD can demonstrate increased behavioral symptoms. Such symptoms impact the PWD and contribute to caregiver stress. Nonetheless, PWD across the severity continuum often respond favorably to music. Thoughtfully designed music-based interventions (MBIs) may offer PWD opportunities to engage in meaningful activity and socialize. However, empirical evidence to support the use of MBIs with this population is very limited. This pilot study advances a line of research to test and refine a randomized clinical trial design and gather preliminary data on intervention effectiveness beyond a single session.

The overall objectives of this quantitative pilot study are to (i) establish a well-refined clinical trial design, procedures, and outcome measures and (ii) obtain preliminary data of enduring effectiveness of a multimodal music therapy intervention for engaging persons with severe dementia (AMUSED) with regards to behavioral symptoms and speech. AMUSED uses live participant-preferred music and progressively layers singing, touch, and rhythmic instrument playing concurrent with participant behavioral responses. This MBI is grounded in the person-centered Clinical Practice Model for PWD, which provides guidelines for adjusting the degree of support and challenge offered to an individual. This Model is also used to enhance treatment fidelity.

This pilot study builds on a feasibility study that field tested logistics and demonstrated feasibility and acceptability of the AMUSED intervention protocol through a randomized cross-over trial design. The researchers refined recruitment, data collection, protocol training, and intervention processes. As in past similar work, the researchers demonstrated positive engagement during music therapy sessions. However, obtaining longer-term measures of treatment effects (i.e., neuropsychiatric inventory, Fitbit actigraphy, pulse oximetry, functional measures) proved impractical and unreliable in the care milieu. The researchers' recent qualitative work with long-term care staff revealed possible solutions to more feasibly measure such outcomes in a long-term care setting. The current pilot study builds on this past feasibility and qualitative work.

In this quantitative pilot study, the investigators will use a randomized clinical trial design to test methods and procedures that will be used in a future larger clinical trial. This will help enhance the rigor and reproducibility of this research. The aims of this pilot study are to: 1) determine whether the clinical trial protocol is feasible for a full-scale trial, 2) select the most appropriate primary outcome measure(s) of behavioral symptoms of dementia, and 3) determine if spontaneous speech offers a useful indicator of music-based intervention effectiveness in persons with severe dementia. Participants will be older adults with severe dementia who live in a long-term care facility. To isolate the effects of the music and obtain an estimate of cluster effects, care facilities will be randomly assigned to either receive music therapy or reading. Both conditions use the same structure, strategies, and dosage, with music being the key difference.

ELIGIBILITY:
PARTICIPANT Inclusion Criteria:

* 65 years or older
* late-onset dementia diagnosis from a physician
* stable at facility long enough to establish residency and routine at the facility (about 2 months prior to start of study)
* English is primary language (for pilot study practicality and ensure straightforward evaluation of our aims)
* Dementia is severe: As in the feasibility study, residents' charted score on the Brief Inventory of Mental Status (BIMS) < 7 will be used and no independent function in community affairs, hobbies, chores, or personal care. The BIMS is a component of the Minimum Data Set (MDS), a federally mandated clinical assessment for all residents in US Medicare and Medicaid certified care facilities. It is completed periodically and interpreted by a licensed health care professional employed by the facility who has completed requisite training on the assessment.

PARTICIPANT Exclusion criteria:

* music therapy recipient
* co-occurring movement disorder
* preexisting cognitive disability
* Milder dementia (BIMS 7+); Persons with more significant cognitive decline could arguably respond differently to the intervention than those with milder dementia, a notion that is supported by past music therapy research with this population.

FACILITIES - Inclusion Criteria:

* Any facility in Kentucky that provides residential care for persons with severe dementia (up to 8 facilities).
* At least 5 residents must enroll to make the best use of our resources.
* At least 1 facility staff member available to help with recruitment and periodic observable data collection
* Can accommodate consistent session days and times between lunch and dinner, 2 times per week for 40 minutes, for 12 weeks.
* Willing to communicate questions, concerns, and changes in safety protocols to the research team.
* Can provide a space appropriate for a small group activity (3-5 residents plus a group leader).
* Can ensure staff support is available for safely transitioning participants to/from sessions at the agreed upon session days and time.
* Can assert that music therapy from a credentialed music therapist (MT-BC) is not offered by the facility, to prevent "double dosing" (music entertainment is ok).

FACILITIES - Exclusion Criteria:

-Does not meet one or more inclusion criteria.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2025-03-12 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Mean Change from Baseline in Dementia Behavior at 12 Weeks | Baseline, end of Week 12
  The Quick Dementia Behavior Observation Scale (QD-BOS) is an 18-item observational measure (est. 3 min. to complete). Section 1 contains the 11 sub-questions from the Neuropsychiatric Inventory-Nursing Home section C "agitation/aggression" and care staff rate the presence or absence of 8 behaviors in the past week (raw score 0-8), the frequency (raw score 1-4) and severity of behaviors (raw score 1-3), total score (frequency x severity, ranges 1-12), and occupational disruptiveness of those behaviors (raw score 0-5; all ranges higher score indicates worse behavior). Section 2 contains 5 questions regarding observed psychosocial well-being in the past week using a 5-point Likert-type scale (item range 1-5), and an optional open-ended item. Section 3 contains 1 question regarding job-related stress in the past week, using a 5-point Likert-type scale (range 1-5). A lower score indicates worse/less desirable behavior. Completed by care staff at baseline and every 4 weeks.

SECONDARY OUTCOMES:
Mean Change from Baseline in Dementia Behavior at 4 Weeks | Baseline, end of Week 4
  The QD-BOS is an 18-item observational measure (est. 3 min. to complete). Section 1 contains the 11 sub-questions from the Neuropsychiatric Inventory-Nursing Home section C "agitation/aggression" and care staff rate the presence or absence of 8 behaviors in the past week (raw score 0-8), the frequency (raw score 1-4) and severity of behaviors (raw score 1-3), total score (frequency x severity, ranges 1-12), and occupational disruptiveness of those behaviors (raw score 0-5; all ranges higher score indicates worse behavior). Section 2 contains 5 questions regarding observed psychosocial well-being in the past week using a 5-point Likert-type scale (item range 1-5), and an optional open-ended item. Section 3 contains 1 question regarding job-related stress in the past week, using a 5-point Likert-type scale (range 1-5). A lower score indicates worse/less desirable behavior. Completed by care staff at baseline and every 4 weeks.
Mean Change from Baseline in Dementia Behavior at 8 Weeks | Baseline, end of Week 8
  The QD-BOS is an 18-item observational measure (est. 3 min. to complete). Section 1 contains the 11 sub-questions from the Neuropsychiatric Inventory-Nursing Home section C "agitation/aggression" and care staff rate the presence or absence of 8 behaviors in the past week (raw score 0-8), the frequency (raw score 1-4) and severity of behaviors (raw score 1-3), total score (frequency x severity, ranges 1-12), and occupational disruptiveness of those behaviors (raw score 0-5; all ranges higher score indicates worse behavior). Section 2 contains 5 questions regarding observed psychosocial well-being in the past week using a 5-point Likert-type scale (item range 1-5), and an optional open-ended item. Section 3 contains 1 question regarding job-related stress in the past week, using a 5-point Likert-type scale (range 1-5). A lower score indicates worse/less desirable behavior. Completed by care staff at baseline and every 4 weeks.
Mean Change from Baseline in Dementia Behavior at 4-Week Follow-Up (16 Weeks) | Baseline, 4-week follow up (week 16; 4 weeks after removal of treatment)
  The QD-BOS is an 18-item observational measure (est. 3 min. to complete). Section 1 contains the 11 sub-questions from the Neuropsychiatric Inventory-Nursing Home section C "agitation/aggression" and care staff rate the presence or absence of 8 behaviors in the past week (raw score 0-8), the frequency (raw score 1-4) and severity of behaviors (raw score 1-3), total score (frequency x severity, ranges 1-12), and occupational disruptiveness of those behaviors (raw score 0-5; all ranges higher score indicates worse behavior). Section 2 contains 5 questions regarding observed psychosocial well-being in the past week using a 5-point Likert-type scale (item range 1-5), and an optional open-ended item. Section 3 contains 1 question regarding job-related stress in the past week, using a 5-point Likert-type scale (range 1-5). A lower score indicates worse/less desirable behavior. Completed by care staff at baseline and every 4 weeks.
Mean Change from Baseline in Language Function at 12 Weeks | Enrollment, end of Week 12
  To evaluate change in Aphasia Quotient (AQ) from the bedside Western Aphasia Battery-Revised (WAB-R), a standardized assessment used to evaluate language abilities in individuals with aphasia. WAB-R has been used with persons with dementia to assess impact of cognitive change on language function. The AQ provides a summary measure of the severity of language impairment based on performance across several language domains, including spontaneous speech, auditory verbal comprehension, repetition, and naming/word finding. Scores range from 0 to 100; A higher AQ score indicates better language function. Administered by masked outcome assessor in person at baseline and end of Week 12.
Mean Change from Baseline in Cognition at 12 Weeks | Enrollment, end of Week 12
  The Severe Impairment Rating Scale (SIRS) is used to evaluate the severity of cognitive and functional impairment in individuals with severe dementia, including memory, orientation, and daily living activities. Scores range from 0 to 52, with higher scores indicating more severe impairment. Administered by masked outcome assessor in person at baseline, end of Week 12, and at 4-week follow-up after removal of treatment.
Mean Change from Baseline in Cognition at 4-Week Follow-Up | Baseline, 4-week follow up (week 16; 4 weeks after removal of treatment)
  The SIRS is used to evaluate the severity of cognitive and functional impairment in individuals with severe dementia, including memory, orientation, and daily living activities. Scores range from 0 to 52, with higher scores indicating more severe impairment. Administered by masked outcome assessor in person at baseline, end of Week 12, and at 4-week follow-up after removal of treatment.

OTHER OUTCOMES:
Mean Change in Spontaneous Speech at Week 4 | Immediately before and immediately after session 8 at week 4
  Spontaneous speech will be administered 1 hour before and 1 hour after session 8, during week 4, by a masked outcome assessor, who will follow a script of simple social responses, picture description task [cookie theft], and animal and vegetable naming. Responses will be audio recorded for lexical feature analysis using standard and AI approaches.
Mean Change in Spontaneous Speech at Week 8 | Immediately before and immediately after session 16 at week 8
  Spontaneous speech will be administered 1 hour before and 1 hour after session 16, during week 8, by a masked outcome assessor, who will follow a script of simple social responses, picture description task [cookie theft], and animal and vegetable naming. Responses will be audio recorded for lexical feature analysis using standard and AI approaches.
Mean Change in Spontaneous Speech at Week 12 | Immediately before and immediately after session 24 at week 12
  Spontaneous speech will be administered 1 hour before and 1 hour after session 24, during week 12, by a masked outcome assessor, who will follow a script of simple social responses, picture description task [cookie theft], and animal and vegetable naming. Responses will be audio recorded for lexical feature analysis using standard and AI approaches.

CONTACTS AND LOCATIONS:
Overall Officials: Alaine E. Reschke-Hernandez, PhD, Principal Investigator — University of Kentucky
Locations (9):
- United States (9):
  - Cedar Ridge Health Campus, Cynthiana, Kentucky
  - Walker's Trail Senior Living, Danville, Kentucky
  - University of Kentucky, Lexington, Kentucky
  - Magnolia Springs Senior Living, Lexington, Kentucky
  - Sayre Christian Village, Lexington, Kentucky
  - The Homeplace at Midway, Midway, Kentucky
  - Windsor Care Center, Mount Sterling, Kentucky
  - Daisy Hill Senior Living, Versailles, Kentucky
  - Thomson-Hood Veterans Center, Wilmore, Kentucky

IPD SHARING:
Plan to Share IPD: Yes
This is a small pilot study. Pilot data for preliminary effect size estimating will not be publicly shared. Researchers may request de-identified data and study materials from the principal investigator.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 6 months after publication. The principal investigator will consider sharing data and study materials prior to that time frame in consultation with the study team.
Access Criteria: The principal investigator will share data, qualitative and quantitative analysis plans, and study materials with other researchers who provide a reasonable rationale for intended use, by email. Requests will be reviewed by the principal investigator Reschke-Hernandez, all co-investigators, and all study team members.

REFERENCES:
- [Background] Weinfurt KP. Clarifying the Meaning of Clinically Meaningful Benefit in Clinical Research: Noticeable Change vs Valuable Change. JAMA. 2019 Dec 24;322(24):2381-2382. doi: 10.1001/jama.2019.18496. No abstract available. PMID 31790549
- [Background] van der Steen JT, Smaling HJ, van der Wouden JC, Bruinsma MS, Scholten RJ, Vink AC. Music-based therapeutic interventions for people with dementia. Cochrane Database Syst Rev. 2018 Jul 23;7(7):CD003477. doi: 10.1002/14651858.CD003477.pub4. PMID 30033623
- [Background] Reschke-Hernandez AE, Tranel D. Strategies to enhance treatment fidelity and music-based intervention reporting in dementia research. Transl Behav Med. 2024 May 24;14(6):353-358. doi: 10.1093/tbm/ibae003. PMID 38334197
- [Background] Reschke-Hernandez, A.E., Ross, M., Davis, H.R., Latham, E.F. and Veblen, N.B. (2023), Multimodal music therapy intervention for engagement and agitation reduction for persons with severe dementia: Study protocol of a pilot randomized cross-over trial. Alzheimer's Dement., 19: e080171. https://doi.org/10.1002/alz.080171
- [Background] Reschke-Hernandez AE, Gfeller K, Oleson J, Tranel D. Music Therapy Increases Social and Emotional Well-Being in Persons With Dementia: A Randomized Clinical Crossover Trial Comparing Singing to Verbal Discussion. J Music Ther. 2023 Oct 7;60(3):314-342. doi: 10.1093/jmt/thad015. PMID 37220880
- [Background] Reschke-Hernández, A. E. (2021). The Clinical Practice Model for Persons with Dementia: Application to music therapy. Music Therapy Perspectives, 39(2), 133-141. https://doi.org/10.1093/mtp/miab006
- [Background] Reschke-Hernández, A. E. (2019). A clinical practice model of music therapy to address psychosocial functioning for persons with dementia: Model development and randomized clinical crossover trial (NCT03643003). Doctoral dissertation, University of Iowa. https://doi.org/10.17077/etd.59oh-y06y
- [Background] Profyri E, Leung P, Huntley J, Orgeta V. Effectiveness of treatments for people living with severe dementia: A systematic review and meta-analysis of randomised controlled clinical trials. Ageing Res Rev. 2022 Dec;82:101758. doi: 10.1016/j.arr.2022.101758. Epub 2022 Oct 13. PMID 36243355
- [Background] Edwards E, St Hillaire-Clarke C, Frankowski DW, Finkelstein R, Cheever T, Chen WG, Onken L, Poremba A, Riddle R, Schloesser D, Burgdorf CE, Wells N, Fleming R, Collins FS. NIH Music-Based Intervention Toolkit: Music-Based Interventions for Brain Disorders of Aging. Neurology. 2023 May 2;100(18):868-878. doi: 10.1212/WNL.0000000000206797. Epub 2023 Jan 13. PMID 36639235
- [Background] Kistin C, Silverstein M. Pilot Studies: A Critical but Potentially Misused Component of Interventional Research. JAMA. 2015 Oct 20;314(15):1561-2. doi: 10.1001/jama.2015.10962. No abstract available. PMID 26501530